CLINICAL TRIAL: NCT04881799
Title: Phentermine/Topiramate in Adolescents With Type 2 Diabetes and Obesity
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEDS-2021-29785
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Phentermine; Topiramate; Qsymia

STUDY DESIGN:
Intervention Model Description: This is a pilot, pragmatic, randomized trial with a 6-month placebo-controlled period followed by a 6-month open label extension investigating the effects of phentermine/topiramate on BMI, insulin sensitivity, and glycemic control compared to placebo plus standard treatment (metformin + insulin) in adolescents with T2D.
  Individuals, when randomized to phentermine/topiramate therapy will initiate treatment at 3.75 mg/23 mg orally once daily in the morning for 14 days. It will then be increased to 7.5 mg/46 mg orally once daily in the morning for 14 days. It will the be increased to 11.25 mg/69 mg orally once daily in the morning for 14 days and finally to 15 mg/92 mg orally once daily in the morning.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants during the first six months of the study will be randomized to receive either phentermine/topiramate or placebo. Neither the participant, care provider, investigator or study team will know whether the participant is receiving phentermine/topiramate or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo-Controlled Period (Placebo Comparator): Participants in this phase of the study will be randomized 1:1 to receive either phentermine/topiramate or placebo.
  Interventions: Drug: Phentermine/Topiramate (Qsymia); Drug: Placebo
- Open Label Extension (Experimental): Participants in this phase of the study will receive open label phentermine/topiramate.
  Interventions: Drug: Phentermine/Topiramate (Qsymia)

INTERVENTIONS:
Drug: Phentermine/Topiramate (Qsymia) — Maximum dose of 15 mg/92 mg orally once daily in the morning. The dose will be titrated to this level (described earlier).
Drug: Placebo — Daily injection
  Arms: Placebo-Controlled Period

SUMMARY:
As the prevalence of obesity rises in the U.S., so does the incidence of pediatric type 2 diabetes (T2D), which is associated with more aggressive disease progression than in adults. From 2002-2012, the incidence of T2D in youth increased by 7% annually in the U.S. Compared to adults. T2D in adolescents is a much more progressive and recalcitrant disease, characterized by more rapid deterioration of β-cell function and earlier incidence of exogenous insulin dependence and diabetes-related comorbidities. A potential factor that drives the rapid progression of adolescent T2D is obesity (body mass index [BMI] >95th percentile. Effective and safe treatments targeting both obesity and β-cell dysfunction are needed for pediatric T2D.

In 2012, the FDA approved the use of Phentermine/Topiramate for the treatment of obesity in adults. This orally-administered medication is available in mid- (phentermine 7.5 mg; topiramate 46 mg) and high- (phentermine 15 mg; topiramate 92 mg) doses, administered once per day. In a meta-analysis, phentermine/topiramate was shown to be one of the most effective obesity medication currently available. A large dose-ranging trial in adults evaluating phentermine and topiramate as monotherapies vs. phentermine/topiramate demonstrated superior efficacy of the combination with an acceptable safety profile.

Results from a large phase III clinical trial demonstrated placebo-subtracted weight loss of >9% with treatment for one year at the top dose. Importantly, a separate trial demonstrated that the treatment effect is durable out to at least two years.41 The most common side effects in these trials were paresthesia, dizziness, dysgeusia, insomnia, constipation, and dry mouth. Improvements were noted in blood pressure, lipids, glucose, insulin, HOMA-IR, C-reactive protein, and adiponectin.

DETAILED DESCRIPTION:
This is a pilot, pragmatic, randomized trial with a 6-month placebo-controlled period followed by a 6-month open-label extension, investigating the effects of phentermine/topiramate on BMI, insulin sensitivity, and glycemic control compared to placebo plus standard treatment (metformin+insulin) in adolescents with T2D. The purpose of this study is to 1) evaluate the effects of phentermine/topiramate vs. placebo+ standard treatment on BMI in adolescents with T2D and obesity and 2) evaluate the effects of phentermine/topiramate vs. placebo + standard treatment on insulin sensitivity and B-cell function in adolescents with T2D and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to </= 20 years at study entry
* Obesity (BMI >/= the 95th percentile for age and sex)
* HgbA1c >/= 6.5% at type 2 diabetes diagnosis
* Negative diabetes auto-antibodies
* English-speaking and Spanish speaking
* For participants of child-bearing potential: when sexually active, agreement to use two forms of highly effective contraception (oral contraceptive pill, IUD, implant, and/or condoms) during study participation

Exclusion Criteria:

* Pregnancy or lactation
* Newly-initiated or change in dose of weight altering medication within past 6 months, including SGLT-2 inhibitors and DPP-IV inhibitors, liraglutide 1.8 mg and exenatide ER.
* Current or recent (< six months prior to enrollment) use of anti-obesity medication(s) defined as orlistat, phentermine, topiramate, combination PHN/TPM, semaglutide, and/or combination naltrexone/bupropion (monotherapy use of naltrexone or bupropion is not an exclusion)
* Current use of sulfonylureas
* Previous metabolic/bariatric surgery
* Current use of a stimulant medication
* History of glaucoma
* Current or recent (< 14 days) use of monoamine oxidase inhibitor or carbonic anhydrase inhibitors
* Known hypersensitivity to sympathomimetic amines
* Any history of treatment with growth hormone
* any history of bulimia nervosa
* Major psychiatric disorder as determined by the local medical monitor
* Unstable and clinically-diagnosed (defined as documented in the medical record, if available) depression or PHQ-9 score of >/= 15
* Any history of active suicide attempt, a "yes" answer to Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) on the "Suicidal Ideation" portion of the C-SSR, or a "yes" to answer to Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS
* History of suicidal ideation or self-harm within the previous 30 days or a "yes" answer to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act, or behavior) on the "Suicidal Behavior" portion of the C-SSRS and the ideation or behavior occurred within the past month.
* Current pregnancy or plans to become pregnant during study participation
* Current tobacco use
* ALT or AST >/= 3 times the upper limit of normal
* Moderate (Child-Pugh score 7-9) or severe (Child-Pugh score 10-15)
* Bicarbonate <18 mmol/L
* Moderate (creatinine clearance [CrCl] greater than or equal to 30 and less than 50 mL/min) or severe (CrCl less than 30 mL/min) renal impairment
* Any history of seizures

  • BP for ages 13 and older of > 130/80 on 3 separate measurements and for age 12 > 95th percentile on 3 separate measurements
* HR ≥120 bpm on 3 separate measurements
* History of structural heart defect or clinically significant arrhythmia
* Diagnosed monogenic obesity
* Any history of cholelithiasis
* Any history of nephrolithiasis
* Clinically diagnosed hyperthyroidism
* Untreated thyroid disorder or TSH below the lower laboratory limit of normal
* Any disorder, unwillingness, or inability, not covered by any other exclusion criteria, which in the investigator's opinion may put the participant at risk

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | 6 Months
  The percent change in body mass index (BMI) from Baseline to Month 6 will be calculated. BMI is defined as a person's weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Bensignor, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The protocol, statistical analysis plan and final study report will be released to other researchers but will not contain identifying information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 10 years after completion of the study

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04881799/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04881799/ICF_001.pdf